CLINICAL TRIAL: NCT06399289
Title: A Phase 3, Open-label, Multicenter, Pharmacokinetics, Efficacy, and Safety Study of a Recombinant Fusion Protein Linking Coagulation Factor IX With Albumin (rIX-FP) in Previously Treated Chinese Subjects With Hemophilia B
Brief Title: Recombinant Fusion Protein Linking Coagulation Factor IX With Albumin (rIX-FP) in Chinese Subjects With Hemophilia B Previously Treated With FIX Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSL654_3004; 2022-002333-34 (EudraCT Number)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Albumins; albutrepenonacog alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rIX-FP (Experimental): Subjects will receive rIX-FP as an intravenous (IV) infusion for a minimum of 50 exposure days (EDs)
  Interventions: Biological: Recombinant fusion protein linking coagulation factor IX with albumin (rIX-FP)

INTERVENTIONS:
Biological: Recombinant fusion protein linking coagulation factor IX with albumin (rIX-FP) — Lyophilized powder for solution for intravenous injection
  Other Names: rIX-FP; CSL654; Idelvion

SUMMARY:
This study will investigate the pharmacokinetics (PK), efficacy, and safety of rIX-FP for the routine prophylaxis of bleeding episodes in male Chinese previously treated patients (PTPs) with hemophilia B (FIX activity of ≤ 2%). In addition to the scheduled rIX-FP prophylaxis regimen, subjects may also receive rIX-FP episodic (on-demand) treatment for breakthrough bleeding episodes and rIX-FP for the prophylaxis and treatment of bleeding in emergency surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* - Male Chinese subjects aged ≤ 70 years
* - Subjects with documented severe or moderately severe hemophilia B (FIX activity of ≤ 2%)
* - Subjects have received FIX products for ≥ 150 exposure days (EDs) (subjects aged ≥ 6 years) or ≥ 50 EDs (subjects aged < 6 years)
* - Subjects have no confirmed prior history of FIX inhibitor formation

Exclusion Criteria:

* - Known hypersensitivity (allergic reaction or anaphylaxis) to any FIX product or hamster protein.
* - Known congenital or acquired coagulation disorder other than congenital FIX deficiency.
* - Currently receiving intravenous (IV) immunomodulating agents such as immunoglobulin or chronic systemic corticosteroid treatment.
* - Currently receiving a long-acting recombinant FIX treatment such as coagulation factor IX (recombinant), Fc fusion protein (Alprolix®).
* - Use of traditional or herbal Chinese medicine(s) with an impact on hemophilia, including coagulation, within 28 days before Day 1 and / or refusal to abstain from these during the study until the end of the subject's participation in the study.

Max Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-07-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incremental recovery (IR) (plasma FIX activity) | Before, and at 30 minutes after the end of, rIX-FP infusion on Day 1
Maximum plasma concentration (Cmax) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1
Terminal elimination half-life (t1/2) of rIX-FP | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1
Area under the concentration-time curve (AUC) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1
  AUC from time zero to the last measurable concentration (plasma FIX activity) (AUC0-last), and AUC from time zero extrapolated to infinity (AUC0-inf).
Clearance (Cl) of rIX-FP | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1
Annualized spontaneous bleeding rate (AsBR) | Up to 18 months
  AsBR for treated bleeding episodes, by prophylaxis regimen and overall
Number of subjects who develop an inhibitor to FIX | Up to 18 months after rIX-FP infusion

SECONDARY OUTCOMES:
Percentage of area under the concentration-time curve extrapolated (%AUCExt) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1 and at Week 26 (Repeat PK)
Area under the first moment versus time curve extrapolated to infinity (AUMC0-∞) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1 and at Week 26 (Repeat PK)
Mean residence time (MRT) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1 and at Week 26 (Repeat PK)
Apparent volume of distribution during the terminal phase (Vz) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1 and at Week 26 (Repeat PK)
Apparent volume of distribution at steady-state (Vss) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1 and at Week 26 (Repeat PK)
Time to reach Cmax (Tmax) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1 and at Week 26 (Repeat PK)
Elimination rate constant (λz) | Before, and up to 336 hours after the end of, rIX-FP infusion on Day 1 and at Week 26 (Repeat PK)
Incremental recovery (IR) (plasma FIX activity) - Repeat PK | Before, and at 30 minutes after the end of, rIX-FP infusion at Week 26
Maximum plasma concentration (Cmax) - Repeat PK | Before, and up to 336 hours after the end of, rIX-FP infusion at Week 26
Terminal elimination half-life (t1/2) of rIX-FP - Repeat PK | Before, and up to 336 hours after the end of, rIX-FP infusion at Week 26
Area under the concentration-time curve (AUC) - Repeat PK | Before, and up to 336 hours after the end of, rIX-FP infusion at Week 26
  AUC from time zero to the last measurable concentration (plasma FIX activity) (AUC0-last), and AUC from time zero extrapolated to infinity (AUC0-inf).
Clearance (Cl) of rIX-FP - Repeat PK | Before, and up to 336 hours after the end of, rIX-FP infusion at Week 26
Annualized bleeding rate (ABR) | Up to 18 months after rIX-FP infusion
  ABR for treated, untreated, and both treated and untreated bleeding episodes (spontaneous bleeding, traumatic bleeding, unknown bleeding, and total bleeding episodes), by prophylaxis regimen and overall
Annualized joint bleeding rate (AjBR) | Up to 18 months after rIX-FP infusion
  AjBR for treated, untreated, and both treated and untreated bleeding episodes, by prophylaxis regimen and overall
Clinical evaluation of hemostatic efficacy for major bleeding episodes | Up to 18 months after rIX-FP infusion
  The investigator will rate the efficacy of the rIX-FP treatment for major bleeding episodes based on a hemostatic efficacy four point rating scale of "excellent, good, moderate or no efficacy", by prophylaxis regimen and overall
Change in target joints | At baseline and up to 18 months after rIX-FP infusion
Consumption of rIX-FP - number of rIX-FP infusions (doses) | Up to 18 months after rIX-FP infusion
  Consumption of rIX-FP expressed as number of rIX-FP infusions (doses), for the prophylaxis regimens, episodic (on-demand) treatment for bleeding episodes (if any), and total (overall) treatment
Consumption of rIX-FP - IU/kg per subject per month | Up to 18 months after rIX-FP infusion
  Consumption of rIX-FP expressed as total amount (IU/kg) per subject per month, for the prophylaxis regimens, episodic (on-demand) treatment for bleeding episodes (if any), and total (overall) treatment
Consumption of rIX-FP - IU/kg per subject per year | Up to 18 months after rIX-FP infusion
  Consumption of rIX-FP expressed as total amount (IU/kg) per subject per year, for the prophylaxis regimens, episodic (on-demand) treatment for bleeding episodes (if any), and total (overall) treatment.
Number of bleeding episodes requiring rIX-FP to achieve hemostasis | Up to 18 months after rIX-FP infusion
  Number of bleeding episodes requiring 1, ≤ 2, or > 2 infusions (doses) of rIX-FP to achieve hemostasis
Percentage of bleeding episodes requiring rIX-FP to achieve hemostasis | Up to 18 months after rIX-FP infusion
  Percentage of bleeding episodes requiring 1, ≤ 2, or > 2 infusions (doses) of rIX-FP to achieve hemostasis
Number of subjects who develop antibodies against rIX-FP | Before, and up to 18 months after, rIX-FP infusion
Number of subjects who develop antibodies against Chinese hamster ovary host cell protein | Before, and up to 18 months after, rIX-FP infusion
The number of subjects with treatment emergent adverse events (TEAEs) related to rIX-FP | Up to 18 months after rIX-FP infusion
The percentage of subjects with treatment emergent adverse events (TEAEs) related to rIX-FP | Up to 18 months after rIX-FP infusion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — CSL Behring
Locations (7):
- China (7):
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - North China University Of Science And Technology Affiliated Hospital, Tangshan, Hebei
  - Jinan Central Hospital, Jinan, Shandong
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.